CLINICAL TRIAL: NCT00816556
Title: A Randomized Controlled Trial to Evaluate the Efficacy of Low Dose Vaginal Estrogens in the Treatment of Atrophic Vaginitis
Brief Title: A Trial to Evaluate the Efficacy of Low Dose Vaginal Estrogens in the Treatment of Atrophic Vaginitis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Funding
Sponsor: Maire Mac Bride (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Sponsor-Investigator, Maire Mac Bride, M.B., B. Ch., Assistant Professor of Medicine, College of Medicine, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 07-008730; UL1TR000135 (NIH)
Record Dates: First submitted 2008-12-30; First posted 2009-01-01 (Estimated); Results first posted 2014-03-28 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-10

CONDITIONS: Atrophic Vaginitis
MeSH Terms: conditions — Atrophic Vaginitis | interventions — Estriol; Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Estriol (Active Comparator): Estriol 10 micrograms added to Vanicream Lite 0.5 grams applied to vaginal introitus daily for two weeks and then twice weekly for 10 weeks
  Interventions: Drug: Estriol
- Estradiol (Active Comparator): Estradiol valerate 10 micrograms added to Vanicream Lite 0.5 grams applied to vaginal introitus daily for two weeks and then twice weekly for 10 weeks
  Interventions: Drug: Estradiol valerate
- Vanicream Lite (Placebo Comparator): Vanicream Lite 0.5 grams applied to vaginal introitus daily for two weeks and then twice weekly for 10 weeks
  Interventions: Drug: Vanicream Lite

INTERVENTIONS:
Drug: Estriol — Estriol 10 micrograms added to Vanicream Lite 0.5 grams applied to vaginal introitus daily for 2 weeks and then twice weekly for 10 weeks.
  Arms: Estriol
Drug: Estradiol valerate — Estradiol valerate 10 micrograms added to Vanicream Lite 0.5 grams applied to vaginal introitus daily for two weeks and then twice weekly for 10 weeks
  Other Names: Delestrogen
  Arms: Estradiol
Drug: Vanicream Lite — Vanicream Lite 0.5 grams applied to vaginal introitus daily for two weeks and then twice weekly for 10 weeks
  Arms: Vanicream Lite

SUMMARY:
Atrophic vaginitis is a common problem that occurs in up to 40% of postmenopausal women. The main symptoms are dryness, itching and burning in and around the vagina. These symptoms in turn can cause pain with intercourse. Other symptoms can include urinary frequency and urinary urgency. These symptoms are caused by the decreasing levels of estrogens in postmenopausal women.

The current treatment options include hormone replacement therapy by mouth and patch and vaginal creams, tablets and rings. The current guideline recommend using hormone therapy at the lowest dose for the shortest time. We are trying to find the lowest effective dose of estrogen cream that helps with symptoms without causing an increase in estrogens in the blood stream.

We want to compare two estrogen creams, estradiol and estriol, each at very low doses, with a placebo cream. Estradiol cream is available on prescription but we want to see how effective it is at one tenth the commonly prescribed dose. Estriol cream is not commonly prescribed and is only available at compounding pharmacies. We want to see if either of these estrogens is effective at one tenth the usual dose. We also want to see if these creams are effective when massaged onto the outer part of the vagina, rather than the usual method of treatment, which is inserting them into the vagina.

DETAILED DESCRIPTION:
This trial will measure the effects of very low doses of estradiol or estriol cream applied to the vaginal introitus for the treatment of atrophic vaginitis, a common condition affecting up to 40% of postmenopausal women. We will conduct a randomized controlled trial with three arms-estradiol, estriol and placebo. The intervention will last for 12 weeks. The outcomes we will be most interested in are the efficacy of the treatments for symptoms of atrophic vaginitis compared to placebo and whether there is any measurable systemic absorption from the locally applied estrogen creams. These outcomes will be measured, primarily, by the use of patient questionnaires and secondarily, clinical examination scores. Safety will be evaluated with serum estrogen concentrations. All measures will be collected at baseline and at the termination of the study. Hormone concentrations will be collected, additionally, at week 2. This trial will answer important questions regarding the impact of very low doses of locally applied estrogens and symptoms of atrophic vaginitis. It will provide information on effect size and validity of outcome measures. It will also give information about whether low doses of estrogen creams, locally applied to the vaginal introitus, result in systemic absorption

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women (no menses for the previous 12 months)
* Dryness, itching or burning in and around the vagina
* Discontinued hormone replacement therapy (either local or systemic) at least 3 months

Exclusion Criteria:

* Known, suspected, or history of cancer of the breast.
* Known, or suspected estrogen dependent neoplasia (ovarian, endometrial).
* Known hypersensitivity to any component of the medications or base creams.
* Active deep vein thrombosis, pulmonary embolism, or history of these conditions.
* Active or recent (within the past year) arterial thromboembolic disease (stroke, myocardial infarct).
* Liver dysfunction or disease with elevation of aspartate aminotransferase (AST)>1.5x upper level of normal (ULN); Normal for females is 8-43 U/L.
* Undiagnosed abnormal genital bleeding.
* Known chronic lichen sclerosis.
* Known, untreated vaginal infection.
* Not had a normal screening mammogram within the last 15 months.
* Hysterectomy without oophorectomy unless 60 years or older.
* Women taking aromatase inhibitors or tamoxifen.
* Hgb <12.0 or >15.5 g/dL
* Urinalysis showing a urinary tract infection (UTI).

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2008-10; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maire B Mac Bride, MB BCh, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Vanicream Lite 0.5 grams applied to vaginal introitus daily for two weeks and then twice weekly for 10 weeks
Period: Overall Study
Arm/Group | Estriol | Estradiol | Placebo
Started | 20 | 21 | 22
Completed | 18 | 19 | 19
Not Completed | 2 | 2 | 3
Not completed — Adverse Event | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Estriol | Estradiol | Placebo | Total
Number analyzed (Participants) | 18 | 19 | 19 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 18 | 19 | 19 | 56
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 19 | 56
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 19 | 19 | 56

OUTCOME MEASURES:

1. Primary Outcome: Change in Vulvovaginal Atrophy Questionnaire (VVAQ) Scores From Baseline to Week 12
Description: The VVAQ consists of three questions asking the participant to rate the severity and how bothersome each of the symptoms of atrophic vaginitis are (dryness, itching, and burning). It is graded 0 through 10. A higher number indicates less severe and less bothersomeness of the symptom, that is, 0= very severe or bothersome, 10= least severe or bothersome.
Time Frame: baseline, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Estriol | Estradiol | Placebo
Number analyzed (Participants) | 18 | 19 | 19
units on a scale
  Dryness Severity | 3.2 (2.3) | 2.0 (3.3) | 2.7 (2.7)
  Dryness Bothersomeness | 2.3 (2.8) | 2.1 (2.7) | 3.6 (3.1)
  Itching Severity | 1.4 (1.6) | 2.6 (2.9) | 1.9 (2.8)
  Itching Bothersomeness | 1.3 (1.6) | 2.6 (3.0) | 1.7 (2.5)
  Burning Severity | 2.1 (2.6) | 1.5 (2.5) | 1.0 (2.9)
  Burning Bothersomeness | 1.9 (2.7) | 1.5 (2.6) | 1.1 (3.1)
Statistical Analysis 1: Comparison: Estriol vs Estradiol vs Placebo; Dryness severity: P-value for the global F-test testing for all treatment arm effects equal; Test type: Superiority or Other; p = 0.42, ANOVA
Statistical Analysis 2: Comparison: Estriol vs Estradiol vs Placebo; Dryness bothersomeness: P-value for the global F-test testing for all treatment arm effects equal; Test type: Superiority or Other; p = 0.22, ANOVA
Statistical Analysis 3: Comparison: Estriol vs Estradiol vs Placebo; Itching severity: P-value for the global F-test testing for all treatment arm effects equal; Test type: Superiority or Other; p = 0.37, ANOVA
Statistical Analysis 4: Comparison: Estriol vs Estradiol vs Placebo; Itching bothersomeness: P-value for the global F-test testing for all treatment arm effects equal; Test type: Superiority or Other; p = 0.27, ANOVA
Statistical Analysis 5: Comparison: Estriol vs Estradiol vs Placebo; Burning severity: P-value for the global F-test testing for all treatment arm effects equal; Test type: Superiority or Other; p = 0.46, ANOVA
Statistical Analysis 6: Comparison: Estriol vs Estradiol vs Placebo; Burning bothersomeness: P-value for the global F-test testing for all treatment arm effects equal; Test type: Superiority or Other; p = 0.67, ANOVA

2. Secondary Outcome: Change in Serum Estrone (E1) Levels Between Baseline, 2 Weeks, and 12 Weeks
Time Frame: baseline, 2 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Estriol | Estradiol | Placebo
Number analyzed (Participants) | 18 | 19 | 19
pg/ml
  Baseline vs. Week 2 | -0.9 (4.6) | -1.6 (3.8) | 0.5 (4.5)
  Baseline vs. Week 12 | 1.0 (4.4) | 1.2 (5.0) | 1.1 (3.5)
  Week 2 vs. Week 12 | 2.2 (5.6) | 1.5 (3.4) | 0.6 (4.8)
Statistical Analysis 1: Comparison: Estriol vs Estradiol vs Placebo; Baseline vs. week 2: P-value for the global F-test testing for all treatment arm effects equal; Test type: Superiority or Other; p = 0.33, ANOVA
Statistical Analysis 2: Comparison: Estriol vs Estradiol vs Placebo; Baseline vs. week 12: P-value for the global F-test testing for all treatment arm effects equal; Test type: Superiority or Other; p = 0.99, ANOVA
Statistical Analysis 3: Comparison: Estriol vs Estradiol vs Placebo; Week 2 vs. week 12: P-value for the global F-test testing for all treatment arm effects equal; Test type: Superiority or Other; p = 0.58, ANOVA

3. Secondary Outcome: Change in Serum Estradiol (E2) Levels Between Baseline, 2 Weeks, and 12 Weeks
Time Frame: baseline, 2 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Estriol | Estradiol | Placebo
Number analyzed (Participants) | 18 | 19 | 19
pg/ml
  Baseline vs. Week 2 | 0.0 (1.1) | -1.7 (3.3) | 0.5 (1.2)
  Baseline vs. Week 12 | -0.4 (3.0) | 0.6 (1.7) | 0.2 (1.6)
  Week 2 vs. Week 12 | -0.3 (2.8) | 1.9 (3.6) | -0.3 (1.1)
Statistical Analysis 1: Comparison: Estriol vs Estradiol vs Placebo; Baseline vs. week 2: P-value for the global F-test testing for all treatment arm effects equal; Test type: Superiority or Other; p = 0.007, ANOVA
Statistical Analysis 2: Comparison: Estriol vs Estradiol vs Placebo; Baseline vs. week 12: P-value for the global F-test testing for all treatment arm effects equal; Test type: Superiority or Other; p = 0.32, ANOVA
Statistical Analysis 3: Comparison: Estriol vs Estradiol vs Placebo; Week 2 vs. week 12: P-value for the global F-test testing for all treatment arm effects equal; Test type: Superiority or Other; p = 0.02, ANOVA

ADVERSE EVENTS:
Time Frame: The study coordinator contacted the participants every 2 weeks and asked the questions on the Adverse Events Stopping Rules. The participant was contacted again at 4 weeks after completion of the study to determine if further side effects had occurred.
Description: Subjects also completed the Symptoms Inventory Questionnaire at baseline, 2, 4, 8, and 12 weeks. If subjects experienced a serious adverse event they were to be withdrawn from the study. These events included elevated blood pressure, a breakdown of vulvar or vaginal skin, or possible allergy to the medication.
Arm/Group | Estriol | Estradiol | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 3/18 | 0/19 | 1/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Estriol (N=18) | Estradiol (N=19) | Placebo (N=19)
Red Bumpy Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal Spotting (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) — The subject on placebo arm experienced at week 4, the subject on estriol arm experienced 4 weeks after completion of study.
Breast tenderness (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No